CLINICAL TRIAL: NCT00562952
Title: Nt-proBNP Guided Prevention of Cardiovascular Events in a Population of Diabetic Patients Without a History of Cardiac Disease
Brief Title: Nt-proBNP Guided Primary Prevention of CV Events in Diabetic Patients
Acronym: PONTIAC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Martin Huelsmann, Doz., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01/07; EK-Nr 391/2007 (Other: Medical University of Vienna)
Record Dates: First submitted 2007-11-23; First posted 2007-11-26 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus; Heart Failure; Coronary Artery Disease
Keywords: Natriuretic peptide; Prognosis; Diabetes; Heart failure; Heart disease
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure; Coronary Artery Disease; Heart Diseases | interventions — Telmisartan; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patient will receive cardiac therapy to decrease NT-proBNP levels. This will be primarily RAAS-Antagonists and Betablocker. Blood pressure will be lowered to target values. A decrease of NT-proBNP is also known form life-style changes. Thus the patient will be educated to be trained
  Interventions: Drug: Telmisartan, Bisoprolol
- 2 (Placebo Comparator): Patients will be followed 2 years. Care will be given by the responsible unit ( Dept.of Endocrinology) as clinical appropriate. Event rates will be obtained. After one year NT-proBNP will be measured.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Telmisartan, Bisoprolol — Dosage will be given dependent on the NT-pro-BNP levels. Up-titration will be performed until values are decreased to 50% or below normal cut-point
  Arms: 1
Drug: placebo — no intervention
  Arms: 2

SUMMARY:
Increased levels of NT-proBNP are known to increase the risk of cardiac events in diabetic patients. The other way around, patients with normal values have an excellent prognosis on short-term. We intend in our study to proof the hypothesis, whether it is possible to decrease NT-proBNP levels by intensified cardiac prevention care We aim those patients, who already have elevated levels, although no history of a cardiac disease. This decrease in NT-proBNP should be translated consequently in a decrease in cardiac events

DETAILED DESCRIPTION:
Patients with diabetes mellitus have a several-fold increased risk for cardiovascular disease (1-3, 16). Early diagnosis of theses diseases might prevent or at least postpone occurence of clinical manifest CAD and CHF. Multifactorial intervention, with a special interest on cardiac disease are proven to be beneficial for diabetic patients (4). Whether all patients benefit from a multi-drug supply including lipid lowering agents or antihypertensive drugs is not known. Thus, special population have to be defined, who profit most. E.g. the STENO- study population (4) consisted of patients with microalbuminuria. Microalbuminuria is known to be a good marker for outcome in this population (5). Consistently to the fact that microalbuminuria is a good marker for long-term outcome, the STENO-Investigators found a long-term benefit (average 7.8 years) for multi-factorial intervention in this special population. We recently found, that Nt-proBNP (Roche) is an excellent short-term predictor of cardiovascular events and death (10 months on average) in diabetics without a history of cardiac disease (6), which is already known for long-term (7-10). Patients above the normal range have a 10 % risk of first occurrence of a cardiac disease or death within short time. The advantage of Nt-BNP as a marker of risk is based on the fact, that it is increased in all cardiac disease dependent on the severity. Our data reveal that Nt-proBNP is superior to most known markers. The limitations of traditional surrogate marker of risk in diabetic patients was recently discussed in a joint statement of the American Heart and Diabetic Associations ( Diabetes Care 2007 Januar).Whether lowering blood pressure or cholesterol is the optimal surrogate for therapeutic success is questionable. The Jikei Heart study (11) nicely shows a comparable decrease in blood pressure in several treatment groups, but a tremendous difference in outcome. The heart failure paradoxon demonstrates, that in this population patients with low blood pressure (12) or low cholesterol (13) are those with worse prognosis. And heart failure is immanent in diabetes. On the other hand a decrease in Nt-proBNP under therapy is known to be an excellent marker of outcome (14). We hypothesize, that including diabetic patients without a history of cardiac disease but increased levels of Nt-BNP will be an excellent short-term risk-population for prevention therapy. And, decreasing Nt-proBNP levels by optimized therapy will be a good marker for success to decrease the risk for future imminent events

Patients will be randomized into two groups:

Group A: Patients will be cared by a cardiologic unit. In accordance to the guidelines investigations will be performed to proof the existence of a manifest cardiac disease. Further on treatment will be tailored to minimize the individual risk profile in accordance to the guidelines (15). The main therapeutic focus will be a decrease in Nt-proBNP to 50% of the value at index time or below normal values. Secondly, a special focus will be set on optimizing anti-hyperglycemic therapy by a diabetologist (treatment to target). Further guideline-recommended medical treatment will be initiated if not yet started (if no contraindication exists all patients will receive oral anti-platelet therapy and lipid lowering medication). After obtained informed consent, patients will be investigated as clinical appropriate.

Performance of echocardiography is mandatory to exclude aortic stenosis and to proof the existence of heart failure- as recommended by the guidelines. Group A:patients will receive scheduled visits monthly to optimize pharmacologic treatment.

After optimization visits will be performed as clinical appropriate. In between patients have the opportunity to contact a responsible person and will be contacted additionally by telephone to proof therapeutic success. As clinical appropriate every visit laboratory sample will be drawn, demographic data, data about diabetic complications, pulse and blood pressure will be taken, to test, whether treating goals are reached (see CRF for details). After one year a scheduled visit is mandatory to obtain laboratory samples, pulse and blood pressure to proof final therapeutic success based on the goal parameter, cholesterol, Nt-pro-BNP, heart rate, blood pressure, HBA1c. Group B patients will be cared by the treating physicians as before. The patient and the physicians will be informed about the results of the investigations. After 1 year the patients receive a scheduled visit, where demographic data, data about diabetic complications, lab samples, ECG, and blood pressure will be taken. Anamnesis about hospitalization and drug prescription will be obtained. If a patient prematurely dies, data will be obtained by the treating physician or other responsible institutions. After two years only data about hospitalization and death will be obtained by telephone contact with the patient or the Melderegister in Group A and B. Observation period: 1 year Cohort: 150 patients in each group

1. Stamler J., Vaqccaro O., Neaton JD., Wentworth D. Diabetes, other risk factors, and 12year mortality for men screened in the multiple risk factor intervention trial Diabetes Care 1993;16:434-44
2. Kannel WB, McGee DL. Diabetes and cardiovascular risk factors: the Framingham study. Circulation 1979;59(1):8-13.
3. Almdal T, Scharling H, Jensen JS, Vestergaard H. The independent effect of type 2 diabetes mellitus on ischemic heart disease, stroke, and death: a population-based study of 13,000 men and women with 20 years of follow-up. Arch Intern Med 2004;164(13):1422-6.
4. Gaede P, Vedel P, Larsen N, Jensen G, Parving HH, Pedersen O. Multifactorial intervention and cardiovascular disease in patients with type 2 diabetes. N Engl J Med 2003;348:383-93
5. Pambianco G., Costacou T., Orchard TJ The prediction of major outcomes of type 1 diabetes: a 12-year prospective evaluation of three separate definitions of the metabolic syndrome and their components and estimated glucose disposal rate: the Pittsburgh Epidemiology of Diabetes Complications Study experience. Diabetes Care 2007;30(5):1248-54
6. Neuhold S, Nt-BNP as a short-term predictor of cardiovascular hospitalization or death in diabetic patients without history of cardiac disease compared to classical risk-factors EASD Meeting 2007 Amsterdam
7. Dawson A; Jeyasslan S; Morris AD; Struthers AD. B-type natriuretic peptide as an alternative way of assessing total cardiovascular risk in patients with diabetes mellitus Am J Cardiol.2005 Oct 1;96(7):933-4
8. Tarnow L; Plasma N-terminal pro-B-type natriuretic peptide and mortality in type 2 diabetes Diabetologia 2006;49: 2256-2262
9. Gaede Hildebrandt P, Hess G, Parving HH, Pedersen O. P; Plasma N-terminal pro-brain natriuretic peptide as a major risk marker for cardiovascular disease in patients with type 2 diabetes and microalbuminuria Diabetologia 2005;48:156-163
10. Bhalla MA; Prognostic role of b-type natriuretic peptide levels in patients with type 2 diabetes mellitus JACC 2004;44:1047-54
11. Mochizuki S, Dahlöf B, Shimizu M, Ikewaki K, Yoshikawa M, Taniguchi I, Ohta M, Yamada T, Ogawa K, Kanae K, Kawai M, Seki S, Okazaki F, Taniguchi M, Yoshida S, Tajima N; Jikei Heart Study group. Valsartan in a Japanese population with hypertension and other cardiovascular disease (Jikei Heart Study): a randomised, open-label, blinded endpoint morbidity-mortality study. Lancet. 2007 Apr 28;369(9571):1431-9.
12. Lee T, Chen J, Cohen D, Tsao L. The association between blood pressure and mortality in patients with heart failure Am Heart J 2006 Jan;151(1):76-83
13. Rauchhaus M, Clark AL, Doehner W, Davos C, Bolger A, Sharma R, Coats AJ, Anker SD. The relationship between cholesterol and survival in patients with chronic heart failure. J Am Coll Cardiol 2003 Dec 3;42(11):1933-40
14. Bettencourt P, Friões F, Azevedo A, Dias P, Pimenta J, Rocha-Gonçalves F, Ferreira A.

    Prognostic information provided by serial measurements of brain natriuretic peptide in heart failure. Int J Cardiol. 2004 Jan;93(1):45-8.
15. Guidelines on diabetes, pre-diabetes, and cardiovascular diseases: executive summary. The Task Force on Diabetes and Cardiovascular Diseases of the European Society of Cardiology (ESC) and of the European Association for the Study of Diabetes (EASD). Eur Heart J. 2007 Jan;28(1):88-136.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Known Diabetes mellitus > 6 months
* Increased Nt-proBNP above 125pg/ml
* Given informed consent

Exclusion Criteria:

* Disease other than diabetes, with a life expectancy below 1 year
* patients who suffer from chronic infection or malignant disease
* Women in childbearing age without contraceptive
* History of cardiac disease
* systemic cortisone treatment
* patients who are on chronic or acute hemodialysis, ultra filtration or peritoneal dialysis

Ages: 19 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Reduction in cardiac events | 2

SECONDARY OUTCOMES:
Decrease in NT-pro-BNP in the treatment arm | 1
Reduction in NT-proBNP | 1

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Huelsmann, MD, Principal Investigator — Medical University of Vienna Dept.of Cardiology; Richard Pacher, MD, Principal Investigator — Medical University of Vienna Dept. of Cardiology; Martin Clodi, MD, Study Director — Medical University of Vienna Dept. of Endocrinology
Locations (2):
- Austria (2):
  - General Hospital of Vienna Department of Endocrinology, Vienna
  - Medical University of Vienna, Vienna

REFERENCES:
- [Derived] Huelsmann M, Neuhold S, Resl M, Strunk G, Brath H, Francesconi C, Adlbrecht C, Prager R, Luger A, Pacher R, Clodi M. PONTIAC (NT-proBNP selected prevention of cardiac events in a population of diabetic patients without a history of cardiac disease): a prospective randomized controlled trial. J Am Coll Cardiol. 2013 Oct 8;62(15):1365-72. doi: 10.1016/j.jacc.2013.05.069. Epub 2013 Jun 27. PMID 23810874